CLINICAL TRIAL: NCT00870506
Title: Community-based Intervention to Enhance Signing of Organ Donor Cards
Brief Title: Community Trial to Enhance Organ Donation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Robert Wood Johnson Foundation (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P60MD002265DT1; 1P60MD002265-01 (NIH)
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Tissue and Organ Procurement; Health Behavior
Keywords: Randomized Controlled Trial; Healthcare Disparities
MeSH Terms: conditions — Health Behavior | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (No Intervention): No intervention (control)
- 1 (Experimental): 5-minute video on donation and transplantation
  Interventions: Behavioral: video

INTERVENTIONS:
Behavioral: video — 5-minute video compared (intervention) to no video and no other intervention (control)
  Arms: 1

SUMMARY:
The purpose of this study is to determine the effect of a 5-minute video intervention regarding organ donation and transplantation on increasing the number of organ donor cards signed in Northeastern Ohio Bureau of Motor Vehicles (OBMV) branches and on willingness to donate organs while living. The investigators hypothesize that persons in the intervention group will sign more donor cards and be more willing to donate organs while living than persons in the control group.

DETAILED DESCRIPTION:
We propose a community-based randomized controlled trial involving 450 intervention and 450 control patrons visiting Ohio Bureau of Motor Vehicle branches (OBMV) to obtain a driver's license. Interventions patrons will watch a 5-minute video prior to entering the OBMV. Study personnel will interview intervention and control patrons after they leave the OBMV to determine whether they signed an organ donor card. We will also determine the effect of the video intervention on willingness to donate organs while living.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Applying for driver's license, driver's permit or state id

Exclusion Criteria:

* Non-English speaking
* Persons who have already signed donor card

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 973 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Proportion of signed donor cards | One day

SECONDARY OUTCOMES:
Proportion of participants willing to donate organs while living | One Day

CONTACTS AND LOCATIONS:
Overall Officials: John D Thornton, MD, MPH, Principal Investigator — Case Western Reserve University
Locations (1):
- Ohio Bureau of Motor Vehicles, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Thornton JD, Alejandro-Rodriguez M, Leon JB, Albert JM, Baldeon EL, De Jesus LM, Gallardo A, Hossain S, Perez EA, Martin JY, Lasalvia S, Wong KA, Allen MD, Robinson M, Heald C, Bowen G, Sehgal AR. Effect of an iPod video intervention on consent to donate organs: a randomized trial. Ann Intern Med. 2012 Apr 3;156(7):483-90. doi: 10.7326/0003-4819-156-7-201204030-00004. PMID 22473435